CLINICAL TRIAL: NCT04200261
Title: Multiple-dose Tolerability and Pharmacokinetic Studies of Benapenem in Clinical Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sihuan Pharmaceutical Holdings Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5081-Ⅰ-1005
Record Dates: First submitted 2019-12-13; First posted 2019-12-16 (Actual); Last update posted 2019-12-16 (Actual); Status verified 2019-07

CONDITIONS: Multiple-dose Tolerability and Pharmacokinetic Studies of Benapenem in Clinical Healthy Subjects
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Banapenem (Experimental): 2000 mg group is performed firstly. After completion of observation and confirming that the drug can be safely tolerated, study on 3000 mg group is then performed
  Interventions: Drug: Banapenem
- placebo (Placebo Comparator): sodium chloride injection Once daily for 7 days
  Interventions: Drug: sodium chloride

INTERVENTIONS:
Drug: Banapenem — 2000 mg group is performed firstly. After completion of observation and confirming that the drug can be safely tolerated, study on 3000 mg group is then performed
  Arms: Banapenem
Drug: sodium chloride — sodium chloride
  Arms: placebo

SUMMARY:
To observe the pharmacokinetic profiles of benapenem and its major metabolites in healthy volunteers after continuous multiple-dose benapenem, providing evidence for phase Ⅱ/Ⅲclinical study.

ELIGIBILITY:
Inclusion Criteria:

* 1、 Male or female healthy subjects, aged 18~45(including 18 and 45 years); 2、Body weight ≥ 50 kg and body mass index 19.0~24.0 kg/m2; 3、Prior to the test, physical examination, blood routine, urine routine, liver and kidney functions, and related examinations normal, or mild abnormalities in indicators while without clinical significance as indicated by the investigator ; 4、Normal or mild abnormalities without clinical significance in the standard 12-lead ECG; 5、 Signing informed consent form.

Exclusion Criteria:

* 1、Having a serious systemic disease, infectious disease or mental disorder; 2、Regular smoking, alcohol abuse, and drug abuse ; 3、Use of drugs known damage to an organ within three months; 4、History of specific allergies, or history of drug allergy, especially those allergic to lactams and excipients of test drug; 5、Febrile illnesses within three days before the screening; 6、Patients with mental illness or psychotic disorder in the past; 7、Past mental and nervous system diseases (epilepsy, stroke, cerebrovascular disorder, etc.), gastrointestinal disorder (such as stomach ulcers, gastritis, etc.) or disorder of other systems (such as cardiovascular, respiratory, hematological, or endocrine system, etc.) diseases or medical history; 8、Habitually taking any medication, including traditional Chinese medicine; 9、Having taken any medication that may affect test results within two weeks before the screening, such as antibiotics, NSAIDs, aluminum- or magnesium-containing antacids, diuretics, anticoagulants, central nervous system depressants, and any drug that may affect the drug absorption; 10、Having participated in other investigational drug trial in the preceding three months; 11、Blood donation for 360 ml or more within three months before the screening; 12、Heart rate < 50 bpm or > 100 bpm; 13、Systolic blood pressure<90mmHg or ≥ 140mmHg, diastolic blood pressure ≥ 90 mmHg or <60mmHg ; 14、Women who are pregnant or breastfeeding, or who may be pregnant without adopting acceptable contraception, or who have a positive result in serum pregnancy test; 15、Women who are planning to become pregnant within 6 months, or male subjects who are planning to make his spouse pregnant within 6 months; 16、HBsAg, HCV antibody, HIV antibody, and Treponema pallidum antibody positive; 17、Urine drug-of-abuse testing positive; 18、Any other factor that makes the subject not suitable for the trial as indicated by the investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Ten men, ten women
Enrollment: 20 (Estimated)
Dates: Start 2019-12-16 (Estimated); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
AUC(0-t) of Benapenem | Pre dose and 0.25,1,1.25,1.5, 2, 3,5,8,12, 24,72,96,120,144,144.5,145,145.25,145.5,146,147,149,152,156,168,180,192hours after first Dosing
  AUC(0-t) is the area under the curve from time 0 to t
Maximum observed plasma concentration (Cmax) of Benapenem | Pre dose and 0.25,1,1.25,1.5, 2, 3,5,8,12, 24,72,96,120,144,144.5,145,145.25,145.5,146,147,149,152,156,168,180,192hours after first Dosing
  Maximum observed plasma concentration (Cmax) of Benapenem in healthy subjects
Time to maximum observed plasma concentration (tmax) of Benapenem | Pre dose and 0.25,1,1.25,1.5, 2, 3,5,8,12, 24,72,96,120,144,144.5,145,145.25,145.5,146,147,149,152,156,168,180,192hours after first Dosing
  Time to maximum observed plasma concentration (tmax) of Benapenem in healthy subjects
Time to elimination half-life (t1/2) of Benapenem | Pre dose and 0.25,1,1.25,1.5, 2, 3,5,8,12, 24,72,96,120,144,144.5,145,145.25,145.5,146,147,149,152,156,168,180,192hours after first Dosing
  Time to elimination half-life (t1/2) of Benapenem in healthy subjects

SECONDARY OUTCOMES:
Number of subjects with clinically significant findings in vital signs | Screening, Day1, Day2, Day3, Day4, Day5, Day6, Day7, Day8, Day9, Day10 after Dosing
  Vitals signs such as systolic and diastolic blood pressure, heart rate, and pulse rate will be measured in a semi-supine position after 5 minutes of rest
Number of subjects with clinically significant findings in laboratory parameters | Screening, Day1, Day2, Day3, Day4, Day5, Day6, Day7, Day8, Day9, Day10 after Dosing
  Hematology and Clinical Chemistry and Urine routine abnormalities will be monitored
Number of subjects with clinically significant 12-lead ECGs | Screening, Day1, Day2, Day4, Day5,Day7, Day8, Day10 after Dosing
  Single 12-lead ECGs will be obtained using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QTcF intervals.
Number of subjects with adverse events and serious adverse events | From Screening to Day 10 after dosing
  All adverse events will be monitored in each group subjects

CONTACTS AND LOCATIONS:
Overall Officials: yuan lv, Doctor, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking university first hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No